CLINICAL TRIAL: NCT01234116
Title: A Prospective, Randomized, Open Label Study to Evaluate the Safety and Tolerability of Raltegravir + Truvada Versus Kaletra + Truvada, for Post-exposure Prophylaxis in Health Care Workers
Brief Title: Post-Exposure Prophylaxis in Health Care Workers
Acronym: PEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Indira Brar, MD, Senior Staff Physician Infectious Disease, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PEP Study; 37384 (Other Grant/Funding Number: Merck Pharmaceuticals)
Record Dates: First submitted 2010-11-02; First posted 2010-11-04 (Estimated); Results first posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: Post exposure prophylaxis; Health Care Workers
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Raltegravir Potassium; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Kaletra (Active Comparator): Arm 1: Kaletra two tabs twice a day + Truvada one pill once a day.
  Interventions: Drug: emtricitabine/tenofovir disoproxil fumarate
- Raltegravir (Active Comparator): Arm 2: Raltegravir 400 mg, one pill twice a day + Truvada one pill once a day.
  Interventions: Drug: emtricitabine/tenofovir disoproxil fumarate

INTERVENTIONS:
Drug: emtricitabine/tenofovir disoproxil fumarate — Each health care worker will receive one of the Treatment Arms for 28 days.
  Other Names: Truvada; Isentress; Kaletra

SUMMARY:
Objective: The objective of this study is to determine the safety and tolerability of Post-exposure Prophylaxis (PEP) with a regimen of Truvada + Kaletra among health care workers (HCWs) at Henry Ford Hospital.

Hypothesis: Raltegravir is safe and better tolerated compared with Kaletra, each in combination with Truvada, as assessed by review of completion rates of PEP and also review of completed safety data.

DETAILED DESCRIPTION:
Health Care Workers that have occupational exposure to blood are at risk for HIV infection. Prevention of blood exposure, through safer practices, barrier precautions, safer needle devices, and other innovations, is the best way to prevent infection with HIV and other bloodborne pathogens.

Though these strategies have been successful in reducing the frequency of blood exposure and needlestick injuries in the past decade, the hazard has not been eliminated. As of December 2001, the CDC had received voluntary reports of 57 documented cases of HIV seroconversion temporally associated with occupational exposure to HIV among U.S. health care personnel. An additional 138 infections among health care personnel were considered possible cases of occupational transmission. Because there is no cure or effective vaccine for HIV, optimal post exposure care, including the administration of antiretroviral drugs to prevent HIV infection, remains a high priority in protecting health care workers.

ELIGIBILITY:
Inclusion Criteria:

* Adult (at least 18 years of age)employees of HFH
* History of occupational exposure to bodily fluids
* Negative HIV test
* The ability to understand a written informed consent form, which must be obtained prior to initiation of any study procedures

Exclusion Criteria:

* Positive pregnancy test
* Females who are breastfeeding
* History of renal disease
* Contraindication for treating patient with components of PEP regimen
* Greater than one dose of PEP medication for this exposure event

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2011-02; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Indira Brar, M.D., Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Kaletra | Raltegravir
Started | 8 | 8
Completed | 4 | 7
Not Completed | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Kaletra | Raltegravir | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 8 | 16
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Evidence of Toxicity. Toxicity Was Measured as Any Adverse Event; Nausea, Vomiting, Diarrhea. Elevated Liver Function Tests.
Description: Descriptive study describing toxicity between the 2 groups
Time Frame: Variables to be measured within 4 weeks between groups.
Measure: Number; unit: adverse events
Arm/Group | Kaletra | Raltegravir
Number analyzed (Participants) | 4 | 7
adverse events | 4 | 4

2. Secondary Outcome: Number of Participants That Were HIV Infected
Description: Any patient that gets HIV infected inspite of receiving PEP will be described
Time Frame: HIV ELISA measured within 24 weeks between groups
Measure: Number; unit: participants
Arm/Group | Kaletra | Raltegravir
Number analyzed (Participants) | 4 | 7
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected for 4 weeks from commencement of PEP regimen
Arm/Group | Kaletra | Raltegravir
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/7
Other Adverse Events (participants affected / at risk) | 4/4 | 4/7
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kaletra (N=4) | Raltegravir (N=7)
other (Gastrointestinal disorders) | 4 (17) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes